CLINICAL TRIAL: NCT04312126
Title: Mechanisms Underlying the Beneficial Effects of Naps on Motor Learning
Brief Title: The Beneficial Effects of Naps on Motor Learning
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200060; 20-N-0060
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08-12

CONDITIONS: Stroke
Keywords: Motor Skill; Sleep; Neural Replay; Natural History
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1: 46 healthy young (18-35) volunteers
- Arm 2: 46 healthy older (50-80) volunteers
- Arm 3: 46 chronic (>6 months post-stroke) stroke patients
  Interventions: Device: MRI system; Device: MEG system

INTERVENTIONS:
Device: MRI system — MRI system - GE Discovery MR750 3T
  Groups: Arm 3
Device: MEG system — MEG system The CTF MEG 275 Magnetoencephalography (MEG) scanner system
  Groups: Arm 3

SUMMARY:
Background:

Memory consolidation is the process by which memories become stable, long-term representations in the brain. Consolidation of a motor skill is dependent upon sleep. Some research shows that daytime naps improve people s motor performance and memory retention. Researchers want to find out how daytime naps may contribute to learning and support consolidation of motor skill memories.

Objective:

To learn the role of memory replay during wakeful rest and sleep (naps) in retaining a newly learned skill.

Eligibility:

English-speaking adults ages 18 and older with chronic stroke, or healthy, right-handed, English-speaking adults ages 18-35 and 50-80

Design:

Participants will be screened with:

* medical history
* neurological history
* medicine review
* medical exam
* neurological exam.

Participants will have a magnetic resonance imaging (MRI) scan of the brain. For this, they will lie down in a scanner. The scanner makes loud noises, so they will wear earplugs. They will fill out an MRI screening form before each MRI.

Participants will also have magnetoencephalography (MEG). MEG maps brain activity. It does this by recording the magnetic fields produced by naturally occurring electrical currents in the brain. For MEG, participants will lie down in the MEG room. Their eye movements may be recorded by a video camera.

Participants will have behavior testing. They will practice typing random keys. Then they will repeatedly type a custom sequence that they see on a computer screen. Then they will take a 2-hour nap. Then they will type the same sequence again.

Participants will have no more than 4 visits at the NIH over 3 months. Visits will last 2-4 hours each.

DETAILED DESCRIPTION:
Study Description:

We will investigate the within-individual contribution of wakeful and sleep neural replay to motor skill consolidation in three groups: (a) young healthy subjects, (b) older healthy subjects and (c) patients with chronic stroke.

Objectives:

The primary aim is to determine the relative contribution of neural replay during wakeful rest and sleep to consolidation of a newly learned skill in young and older healthy volunteers, and in chronic stroke patients with magnetoencephalography (MEG). The secondary aim is to evaluate differences in replay rates between these subject cohorts. We will also explore differences in replay rates, spatiotemporal dynamics of neural replay and sleep spindles to generate additional hypotheses and preliminary data for future studies.

Endpoints:

The primary endpoint measure is motor skill consolidation (i.e., offline change in correct sequence typing speed following a nap). The secondary endpoint measure is neural replay rate. Exploratory endpoints measures are spatial (i.e. - parcellated source space) and time-frequency maps of neural replay during wakeful rest and sleep, and changes in button-press finger movement kinematics during learning.

ELIGIBILITY:
* HEALTHY VOLUNTEERS:

INCLUSION CRITERIA:

* Age 18-35 (Arm 1) or 50-80 (Arms 2).
* English speaking.
* Clear right-hand dominance (>74 on Edinburgh Handedness Inventory).
* Normal neurological examination as determined by the screening clinician.

EXCLUSION CRITERIA:

* HCPS affiliated NIH staff (i.e. - staff from our section).
* Current pregnancy.
* Contraindications for MRI or MEG.
* Use of sleep medications within 24 hours of Experimental Session participation.
* Severe or progressive neurological, psychological or medical condition as determined by the screening clinician.

STROKE PATIENTS:

INCLUSION CRITERIA:

* Age 18 or older
* Willing and able to provide consent
* Experienced a stroke 6 months ago or more that affected at least one of the upper extremities at time of stroke diagnosis
* Ability to perform the study task as assessed during physical examination
* English-speaking

EXCLUSION CRITERIA:

* HCPS-affiliated NIH staff (i.e. - staff from our section).
* Current pregnancy
* History of large stroke lesions in brainstem or cerebellum as determined by screening clinician
* Severe or progressive neurological disorder other than stroke (e.g., Parkinson s disease or multiple sclerosis) as determined by the screening clinician
* Uncontrolled heart, lung, kidney, gastrointestinal, metabolic, psychiatric, sleep, or endocrine disorders as determined by the screening clinician
* Contraindications for MRI or MEG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Right-handed adults between the ages of 18 and 80.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint measure is the degree to which motor skill consolidation (i.e., offline change in correct sequence typing speed) is predicted by replay rates during wakeful rest and sleep, and spindle rates during sleep (i.e. multiple r... | 4 years
  The primary endpoint measure is the degree to which motor skill consolidation (i.e., offline change in correct sequence typing speed) is predicted by replay rates during wakeful rest and sleep, and spindle rates during sleep (i.e. multiple regression model with 3 predictors).

SECONDARY OUTCOMES:
Exploratory endpoints measures are spatial (i.e. - parcellated source space) and time-frequency maps of neural replay during wakeful rest and sleep. | 4 years
  Exploratory endpoints measures are spatial (i.e. - parcellated source space) and time-frequency maps of neural replay during wakeful rest and sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-N-0060.html